CLINICAL TRIAL: NCT05391633
Title: Effect of Recorded Maternal Voice on Quantitative EEG (qEEG) as a Marker for Developmental Risk in the Preterm Newborn
Brief Title: Maternal Voice and Quantitative EEG (qEEG)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Per PI, enrollment stopped due to a lack of continued funding and staffing
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Aaron Cardon, Assistant Professor of Neurology, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 21-417
Record Dates: First submitted 2022-02-15; First posted 2022-05-26 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Prematurity; Development Delay; Premature Birth
Keywords: quantitative EEG; Spectral Density Analysis; At Risk for Cognitive Delay; Premature Birth 28-32 weeks gestation
MeSH Terms: conditions — Premature Birth; Learning Disabilities

STUDY DESIGN:
Intervention Model Description: Crossed design, between-group and within-group pre- and post-intervention changes in primary variable.
Who Masked: Investigator, Outcomes Assessor
Masking Description: NICU Investigator will provide the intervention versus placebo, with subject identification unlinked to randomization status. EEG reader, qEEG pruner and qEEG analyst will remain blinded to subject allocation until all data is extracted from each subject's EEG and medical record. To further prevent bias, group assignment unidentified as to control versus intervention will be maintained until all statistical analysis is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Starting at 33 0/7 weeks corrected gestational age (regardless of birth gestation), infants randomized to the non-intervention arm will be played a blank recording of approximately 60 minutes duration, once every 24 hours for a 2-week (14 day) period.
  Interventions: Behavioral: Placebo Recording
- Recorded Voice Exposure (Experimental): Starting at 33 0/7 weeks corrected gestational age (regardless of birth gestation), infants randomized to the intervention arm will be played a recording of their mother's voice with approximately 60 minutes of scripted content, once per 24 hours for a 2-week (14 day) intervention period. (Mothers will be recorded reading a children's book and the recording will be looped to create the 60 minutes of content).
  Interventions: Behavioral: Recorded Maternal Voice

INTERVENTIONS:
Behavioral: Recorded Maternal Voice — 60-minute looped recording of maternal voice, played once daily for 14 total days.
  Arms: Recorded Voice Exposure
Behavioral: Placebo Recording — 60-minute blank recording played once daily for 14 total days.
  Arms: Placebo

SUMMARY:
A short-term randomized, blinded placebo-controlled trial, in premature infants in the neonatal intensive care unit (NICU) at 33-35 weeks post-conceptional age, of recorded maternal voice on quantitative EEG (spectral power density) as a marker of development.

DETAILED DESCRIPTION:
This will be a randomized placebo-controlled clinical trial. Infants consented to participate will be randomized into the intervention arm or non-intervention arm by sealed unmarked envelope.

All consented participants will have an initial EEG of 60-90 minutes duration, performed at 32 5/7 - 32 6/7 weeks (and after 72 hours of life).

Starting at 33 0/7 weeks corrected gestational age (regardless of birth gestation), eligible subjects will proceed with randomized intervention or placebo for a 2-week (14 day) intervention period.

All infants will receive a 2nd EEG of 30-60 minutes duration, performed between 35 0/7 - 35 6/7 weeks corrected gestational age, following completion of either the intervention or non-intervention arm (with the goal of the 2nd EEG occurring within 48 hours of infants having completed the intervention vs. non-intervention arm).

EEG technician and all persons reviewing, pruning and analyzing data from the qEEG will be blinded to whether the infant was in the intervention or the non-intervention arm.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at 28 0/7 - 32 3/7 weeks gestation (to allow for infants born at 32 3/7 weeks to have initial EEG performed after 72 hours of life and prior to initiating intervention or non-intervention arm at 33 0/7 weeks gestation)
* Mother available to provide voice recording, and have ability to converse and read in English (as the scripted content for the intervention will be provided in English)

Exclusion Criteria:

* Infant with Critical Congenital Cardiac Disease
* Infant with Chromosomal anomaly or Inborn Error of Metabolism
* Infant with known Neurologic disorder/abnormality - including hypoxic-ischemic encephalopathy (HIE), intraventricular hemorrhage (IVH), periventricular leukomalacia (PVL), seizure activity, anatomic abnormality
* Infant receiving antiepileptic or sedation medications prior to EEG
* Initial EEG abnormal with epileptiform activity or not consistent with corrected gestational age
* Mother not available to provide voice recording in English
* Unable to obtain consent from mother due to maternal health issues following delivery (such as mother requiring intubation or sedation following delivery
* Mothers who are prisoners (as the study team would like to have continuing communication during the study period as needed)
* Mothers who are <18 years of age will not be approached for consent
* Any mother that is not able to consent due to having a legal representative will not be approached for consent
* Any infant that is planned to be placed for adoption, is in foster care or is a ward of the state

Ages: 28 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-06-12 (Actual)

PRIMARY OUTCOMES:
qEEG change: within | 2 weeks
  Change in relative spectral power, within group, of alpha (8-13 Hz) and beta (14-20 Hz) band
qEEG change: between | 2 weeks
  Difference in relative spectral power, between groups, of alpha (8-13 Hz) and beta (14-20 Hz) band, at baseline and post-treatment

SECONDARY OUTCOMES:
Time to hospital discharge (between groups) | Approximately 7-10 weeks, at NICU discharge date which typically occures around post-conceptional age 39-42 weeks.
  Birth Date to NICU discharge Date
Feeding | Approximately 7-10 weeks, at NICU discharge date which typically occures around post-conceptional age 39-42 weeks.
  Time to full nippled feeds prior to discharge (between groups), gathered retrospectively by chart review at NICU discharge date.
NEC/Sepsis | Approximately 7-10 weeks, at NICU discharge date which typically occures around post-conceptional age 39-42 weeks.
  Episodes of necrotizing enterocolitis (NEC) and/or Sepsis (between groups), gathered retrospectively by chart review at NICU discharge date.
Duration of O2 support | Approximately 7-10 weeks, at NICU discharge date which typically occures around post-conceptional age 39-42 weeks.
  Duration of supplemental O2 needs (between groups), gathered retrospectively by chart review at NICU discharge date.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Cardon, MD, Study Chair — University of New Mexico, Health Sciences Center; Dawn Novak, MD, Principal Investigator — University of New Mexico, Health Sciences Center; Meghan Groghan, Study Director — University of New Mexico, Health Sciences Center
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No